CLINICAL TRIAL: NCT05863377
Title: The Efficacy of Chemotherapy Alone in Patients With Poor-differentiated Early-stage Cervical Cancer But Without the Criteria for Adjuvant Radiotherapy According to NCCN Guidelines
Brief Title: Efficacy of Chemotherapy Alone in Patients With Poor-differentiated Early-stage Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-197
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-01

CONDITIONS: Cervical Cancer
Keywords: early-stage; chemotherapy alone; poor differentiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjuvant Chemotherapy Group: The patients of this group receive adjuvant chemotherapy after surgery.
- No-Further Treatment Group: The patients of this group only receive regular follow-up without adjuvant therapy.

SUMMARY:
This study is aimed to enroll patients with early-stage cervical cancer (FIGO 2018 IB1-IB2) who undergo radical hysterectomy and the postoperative pathology doesn't meet Sedlis criteria or the "four-factor" model but with poorly differentiated squamous/adenocarcinoma/adenosquamous carcinoma. Patients will be randomly divided into two groups in a 1:1 ratio. The experimental group received 4 courses of paclitaxel and cisplatin (once every 3 weeks) for adjuvant chemotherapy within 4 weeks after surgery, while the control group don't not receive any adjuvant therapy but only received regular follow-up. The disease status of all patients will be evaluated within 4 weeks after the end of all treatment and every 12 weeks thereafter, including gynecological examination, laboratory indicators, imaging evaluation, and the prognosis of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. The age of patients is 18-70 years old.
2. Patients with cervical cancer who undergo radical hysterectomy and pelvic lymphadenectomy as initial treatment (including laparoscopic and abdominal surgery).
3. Clinical stage is IB1-IB2 according to FIGO 2018 stage.
4. The postoperative pathological type is squamous cell carcinoma/adenocarcinoma/adenosquamous carcinoma.
5. The degree of tumor differentiation is poorly differentiated.
6. Do not meet the Sedlis criteria or the four-factor model, but meet one of the following factors: ① LVSI (+); ② tumor diameter > 2cm; ③ Depth of cervical stromal invasion > superficial 1/3; (4) adenocarcinoma.

Exclusion Criteria:

1. Postoperative pathological stage ≥IIA (according to the 2018 FIGO staging system).
2. Patients with the following high risk factors: ① lymph node metastasis; ② parametrial involvement; ③ positive surgical margin; ④ vaginal involvement.
3. Patients received neoadjuvant chemotherapy.
4. There was evidence of distant metastasis on preoperative imaging examination.
5. Patients received postoperative radiotherapy.
6. History of abdominal or pelvic radiotherapy.
7. Patients with other malignant tumors.
8. Patients with missing or partially missing clinical, surgical, and pathological data were lost to follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage (FIGO 2018 IB1-IB2 stage) poorly differentiated cervical cancer diagnosed with radical surgery
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 5 years
  The time between surgery and clinical recurrence.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  The time interval between the cancer diagnosis and the death of any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen Universit, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paik ES, Lim MC, Kim MH, Kim YH, Song ES, Seong SJ, Suh DH, Lee JM, Lee C, Choi CH. Prognostic Model for Survival and Recurrence in Patients with Early-Stage Cervical Cancer: A Korean Gynecologic Oncology Group Study (KGOG 1028). Cancer Res Treat. 2020 Jan;52(1):320-333. doi: 10.4143/crt.2019.124. Epub 2019 Aug 5. PMID 31401822
- [Background] Rotman M, Sedlis A, Piedmonte MR, Bundy B, Lentz SS, Muderspach LI, Zaino RJ. A phase III randomized trial of postoperative pelvic irradiation in Stage IB cervical carcinoma with poor prognostic features: follow-up of a gynecologic oncology group study. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):169-76. doi: 10.1016/j.ijrobp.2005.10.019. Epub 2006 Jan 19. PMID 16427212
- [Background] Rose PG, Ali S, Watkins E, Thigpen JT, Deppe G, Clarke-Pearson DL, Insalaco S; Gynecologic Oncology Group. Long-term follow-up of a randomized trial comparing concurrent single agent cisplatin, cisplatin-based combination chemotherapy, or hydroxyurea during pelvic irradiation for locally advanced cervical cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Jul 1;25(19):2804-10. doi: 10.1200/JCO.2006.09.4532. Epub 2007 May 14. PMID 17502627
- [Background] Ryu SY, Kim MH, Nam BH, Lee TS, Song ES, Park CY, Kim JW, Kim YB, Ryu HS, Park SY, Kim KT, Cho CH, Lee C, Kim SM, Kim BG, Bae DS, Kim YT, Nam JH. Intermediate-risk grouping of cervical cancer patients treated with radical hysterectomy: a Korean Gynecologic Oncology Group study. Br J Cancer. 2014 Jan 21;110(2):278-85. doi: 10.1038/bjc.2013.716. Epub 2013 Dec 19. PMID 24357798
- [Background] Matsuo K, Mandelbaum RS, Machida H, Purushotham S, Grubbs BH, Roman LD, Wright JD. Association of tumor differentiation grade and survival of women with squamous cell carcinoma of the uterine cervix. J Gynecol Oncol. 2018 Nov;29(6):e91. doi: 10.3802/jgo.2018.29.e91. PMID 30207099
- [Background] Rogers L, Siu SS, Luesley D, Bryant A, Dickinson HO. Radiotherapy and chemoradiation after surgery for early cervical cancer. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD007583. doi: 10.1002/14651858.CD007583.pub3. PMID 22592722
- [Background] Sehouli J, Runnebaum IB, Fotopoulou C, Blohmer U, Belau A, Leber H, Hanker LC, Hartmann W, Richter R, Keyver-Paik MD, Oberhoff C, Heinrich G, du Bois A, Olbrich C, Simon E, Friese K, Kimmig R, Boehmer D, Lichtenegger W, Kuemmel S. A randomized phase III adjuvant study in high-risk cervical cancer: simultaneous radiochemotherapy with cisplatin (S-RC) versus systemic paclitaxel and carboplatin followed by percutaneous radiation (PC-R): a NOGGO-AGO Intergroup Study. Ann Oncol. 2012 Sep;23(9):2259-2264. doi: 10.1093/annonc/mdr628. Epub 2012 Feb 21. PMID 22357252
- [Background] Curtin JP, Hoskins WJ, Venkatraman ES, Almadrones L, Podratz KC, Long H, Teneriello M, Averette HA, Sevin BU. Adjuvant chemotherapy versus chemotherapy plus pelvic irradiation for high-risk cervical cancer patients after radical hysterectomy and pelvic lymphadenectomy (RH-PLND): a randomized phase III trial. Gynecol Oncol. 1996 Apr;61(1):3-10. doi: 10.1006/gyno.1996.0087. PMID 8626113
- [Background] Ryu SY, Park SI, Nam BH, Cho CK, Kim K, Kim BJ, Kim MH, Choi SC, Lee ED, Lee KH. Is adjuvant chemoradiotherapy overtreatment in cervical cancer patients with intermediate risk factors? Int J Radiat Oncol Biol Phys. 2011 Mar 1;79(3):794-9. doi: 10.1016/j.ijrobp.2009.11.019. Epub 2010 Apr 24. PMID 20421158